CLINICAL TRIAL: NCT05031065
Title: Identifying Prognostic Indicators for the Development of Radiation-induced Breast Fibrosis
Brief Title: Prognostic Indicators for Radiation-induced Breast Fibrosis
Status: Terminated | Type: Observational
Why Stopped: Loss of Funding
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-0026
Record Dates: First submitted 2021-08-25; First posted 2021-09-01 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women undergoing radiation treatment after lumpectomy for breast cancer.: There is no specific study intervention being used. Samples will be collected from participants undergoing standard of care radiotherapy at pre-specified timepoints.
  Interventions: Radiation: Breast Cancer Radiotherapy

INTERVENTIONS:
Radiation: Breast Cancer Radiotherapy — 4000-4250 cGy in 15-16 daily fractions

SUMMARY:
To study the inflammatory response during and after radiotherapy, especially by measuring the concentration of an enzyme called autotaxin and its product LPA in the blood plasma.

DETAILED DESCRIPTION:
To study the inflammatory response during and after radiotherapy, especially by measuring the concentration of an enzyme called autotaxin and its product LPA in the blood plasma. Autotaxin and LPA cause fibrosis in other situation, but they have not been tested in radiation-induced fibrosis. We will determine if the duration and magnitude of the autotaxin and LPA responses are prognostic for the 15-28% of patients who will develop fibrosis. This fibrosis will be detected by ultrasound and a novel application of elastography, which should provide much earlier and quantifiable fibrotic changes compared to conventional physical examination.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants capable of giving informed consent, or if appropriate, participants having an acceptable individual capable of giving consent on the participant's behalf
2. Age 40 and above.
3. Treatment with breast conserving surgery.
4. Intended adjuvant whole breast radiotherapy dose to a dose of 40-42.5 Gy in 15-16 fractions.
5. Luminal A subtype as determined by clinipathologic factors (ER/PR positive, Her-2 negative, low Ki-67 or low OncotypeDx recurrence score

Exclusion Criteria:

1. Women who have smoked within the last 5 years
2. Patients requiring adjuvant chemotherapy.
3. Requirement for regional nodal radiotherapy.
4. Requirement for tumour bed boost.
5. Breast implants
6. Patients to be treated with partial breast irradiation.
7. Uncontrolled intercurrent illness or active infection.
8. Patients who have previously received chemotherapy.
9. Patients who have previously received chemotherapy.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Born as genetic females
Study Population: We will study a low risk group of 27 post-menopausal patients with luminal A breast cancer after they have received breast conserving surgery (lumpectomy). Women who have smoked or received chemotherapy will be excluded to minimize variables.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Measurement of the ATX-LPA (ATX) inflammatory response to standard RT for breast cancer as a prognostic marker for RT-induced fibrosis. | Samples will be collected four times during RT treatment (3-4 weeks) and once every 3 months for an year.
  Measurement of longitudinal changes in plasma ATX in the irradiated breast.
Measurement of the ATX-LPA-inflammatory (LPA) response to standard RT for breast cancer as a prognostic marker for RT-induced fibrosis. | Samples will be collected four times during RT treatment (3-4 weeks) and once every 3 months for an year.
  Measurement of longitudinal changes in plasma LPA in the irradiated breast.
Measurement of the ATX-LPA-inflammatory (cytokines) response to standard RT for breast cancer as a prognostic marker for RT-induced fibrosis. | Samples will be collected four times during RT treatment (3-4 weeks) and once every 3 months for an year.
  Measurement of longitudinal changes in plasma cytokines in the irradiated breast.
Measurement of the ATX-LPA-inflammatory (chemokines) response to standard RT for breast cancer as a prognostic marker for RT-induced fibrosis. | Samples will be collected four times during RT treatment (3-4 weeks) and once every 3 months for an year.
  Measurement of longitudinal changes in plasma chemokines in the irradiated breast.

SECONDARY OUTCOMES:
Structural changes in the irradiated breast and the non-irradiated breast | 3, 6, 12, 24 and 48 months after RT
  The ultrasound procedure will provide a 3D analysis of the breast structure as well as a measurement of breast elasticity. Fibrotic changes in the breast will be measured by combining the 3D analysis and breast elasticity indices (median (kPa), IQR (kPA) and IQR/median (%))
Acute Radiotherapy Toxicity | Throughout the duration of the study, a total of 4 years .
  Radiotherapy associated toxicities will be assessed per CTCAE v5.0 by the study investigators.
Relationship with Cytomegalovirus infection | Seropositivity for CMV will be checked only at baseline.
  There is evidence that being infected with Cytomegalovirus is likely to increase the response of the autotaxin-lysophosphatidates inflammatory cycle in response to radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Zsolt Gabos, MD, Principal Investigator — AHS-CCI
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided